CLINICAL TRIAL: NCT05096871
Title: Association of Brain Derived Neurotrophic Factor (BDNF) rs6265 Gene Polymorphism With Susceptibility to Epilepsy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Salma Khalaf Abdelmageed, demonstrator of Medical Biochemistry, Sohag University
Other Study IDs: Soh-Med-21-10-18
Record Dates: First submitted 2021-10-14; First posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Epilepsy
Keywords: BDNF in epileptic patients
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: patients with epilepsy
  Interventions: Genetic: Genotyping by Real Time PCR
- Group II: apparently healthy controls with no chronic illness of matched age and sex
  Interventions: Genetic: Genotyping by Real Time PCR

INTERVENTIONS:
Genetic: Genotyping by Real Time PCR — 3 mL of blood will be withdrawn by venipuncture in EDTA tube. DNA extraction will be done after centrifugation and used for genotyping assay of ( BDNF ) gene with the Real- time polymerase chain reaction.
  BDNF level in serum will also be analyzed by Sandwich enzyme linked immunosorbant assay kit ( ELISA).

SUMMARY:
Epilepsy is a common neurological condition that affects people of all ages.Recent studies found that epilepsy is associated with several chromosomal regions, where mutations in these regions cause neurological dysfunction.

BDNF which is the most ample neurotropic factor in the CNS, has survival and growth promoting roles in a variety of neurons. It has been shown to promote excitatory (glutamatergic) synapses while weakening inhibitory (GABAergic) ones.

A nonsynonymous G to A single-nucleotide polymorphism (SNP) exists at position 196 of exon 2 (rs6265), which results in valine (val) to methionine (met) substitution. This polymorphism affects intracellular packaging of pro-BDNF, its axonal transport and in turn, activity-dependent secretion of BDNF at the synapse.

DETAILED DESCRIPTION:
Epilepsy was defined as the separate occurrence of two or more unprovoked seizures, manifested by involuntary motor, sensory, or autonomic, alone or in combination, and not diagnosed as neonatal or febrile seizures. Despite extensive studies, the molecular causes of the disease are not yet discovered completely. A functional imbalance between excitatory (transmitted by glutamate) and inhibitory signals (transmitted by γ-amino butyric acid or GABA) in neural cells has been regarded as a putative contributing factor in epilepsy.

The brain-derived neurotropic factor (BDNF) encodes a small dimeric protein which is the most ample neurotropic factor in the CNS.It has been shown to promote excitatory (glutamatergic) synapses while weakening inhibitory (GABAergic) ones.Any interference with the BDNF signaling pathway may negatively affect downstream neuronal functions and cause neuronal diseases.

A nonsynonymous G to A single-nucleotide polymorphism (SNP) exists at position 196 of exon 2 (rs6265), which results in valine (val) to methionine (met) substitution at codon 66 (val66met), changing the 5' proregion of the human BDNF protein. This polymorphism affects intracellular packaging of pro-BDNF, its axonal transport and in turn, activity-dependent secretion of BDNF at the synapse

ELIGIBILITY:
Inclusion Criteria:

• Epileptic patients aged more than 1 year and less than 15 year who recently had seizures over a period of one year

Exclusion Criteria:

* Patients > 15 years old or less than 1 year.
* Patients that have epilepsy as a result of head injuries, brain tumors , exposure to low oxygen during birth or infections such as meningitis or encephalitis .
* Patients that have no sufficient medical records or unreliable seizure frequency,
* patients with developmental disorders such as Autism and Neurofibromatosis

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients with epilepsy aged from 1 year to less than 15 years, in Pediatric department of Sohag University Hospital and healthy control children of matched age and sex
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Iinvestigate the possible association between BDNF rs6265 polymorphism and epilepsy susceptibility in Egyptian patients | within 3 days after collection of samples
  Genotyping assay of ( BDNF ) rs6265 gene polymorphism by the Real- time polymerase chain reaction.

SECONDARY OUTCOMES:
Assess the utility of serum BDNF concentration as a diagnostic tool for Epilepsy and evaluate its relationship with disease severity | within 3 days after collection of samples
  Measurement BDNF level in serum by Sandwich enzyme linked immunosorbant assay kit

REFERENCES:
- [Background] Egan MF, Kojima M, Callicott JH, Goldberg TE, Kolachana BS, Bertolino A, Zaitsev E, Gold B, Goldman D, Dean M, Lu B, Weinberger DR. The BDNF val66met polymorphism affects activity-dependent secretion of BDNF and human memory and hippocampal function. Cell. 2003 Jan 24;112(2):257-69. doi: 10.1016/s0092-8674(03)00035-7. PMID 12553913
- [Background] Chen ZY, Patel PD, Sant G, Meng CX, Teng KK, Hempstead BL, Lee FS. Variant brain-derived neurotrophic factor (BDNF) (Met66) alters the intracellular trafficking and activity-dependent secretion of wild-type BDNF in neurosecretory cells and cortical neurons. J Neurosci. 2004 May 5;24(18):4401-11. doi: 10.1523/JNEUROSCI.0348-04.2004. PMID 15128854
- [Background] Fisher RS, Acevedo C, Arzimanoglou A, Bogacz A, Cross JH, Elger CE, Engel J Jr, Forsgren L, French JA, Glynn M, Hesdorffer DC, Lee BI, Mathern GW, Moshe SL, Perucca E, Scheffer IE, Tomson T, Watanabe M, Wiebe S. ILAE official report: a practical clinical definition of epilepsy. Epilepsia. 2014 Apr;55(4):475-82. doi: 10.1111/epi.12550. Epub 2014 Apr 14. PMID 24730690
- [Background] Loscher W, Potschka H, Sisodiya SM, Vezzani A. Drug Resistance in Epilepsy: Clinical Impact, Potential Mechanisms, and New Innovative Treatment Options. Pharmacol Rev. 2020 Jul;72(3):606-638. doi: 10.1124/pr.120.019539. PMID 32540959